CLINICAL TRIAL: NCT05036967
Title: HEArt Failure Treatment Patterns: A Descriptive Study in COlombia
Brief Title: A Study to Observe Treatment Patterns in Patients in Colombia Who Have Heart Failure
Acronym: HEATCO
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 21798
Record Dates: First submitted 2021-07-19; First posted 2021-09-08 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Heart Failure (HF) patients: Patients diagnosed with incident HF, in an outpatient setting in Colombia during the time period of 01 JUN 2019 to 31 MAY 2020
  Interventions: Drug: HF medication

INTERVENTIONS:
Drug: HF medication — Treatment initiation patterns of patients with Heart Failure (HF) in an outpatient setting from Colombia.

SUMMARY:
Researchers want to learn more about the treatments doctors choose to treat heart failure.

Heart failure means the heart isn't pumping as well as it should be. Heart failure can lead to other serious medical conditions, and it can lead to hospitalization or death.

There are different types of treatments available for people who have heart failure, and these work in different ways. In this study, the researchers will collect information about Colombian patients who have heart failure.

The main purpose of this study is to identify patterns in the treatments that doctors first prescribe to heart failure patients in Columbia. To do this, the researchers will review information from the patients' medical records and from a drug-dispensing database.

The study will include adult patients who have been diagnosed with heart failure in Columbia from June 1st, 2019 to May 31st, 2020.

There will be no required visits, treatments, or procedures in this study. The researchers will collect information about the treatments the patients have been prescribed by their own doctors.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (older than 18 years) with a diagnosis of HF according to ICD-10 with a dispensing of some medicine and it is registered in the database of Audifarma S.A. during the observation period will be included

Exclusion Criteria:

* Patients with Acute HF without prior diagnosis of HF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with incident HF, in an outpatient setting in Colombia during the time period of 01 JUN 2019 to 31 MAY 2020.
  The universe of the study corresponds to all individuals who are identified in the database as having HF diagnosed by ICD-10 code in the prescription; the target population corresponds to subjects who were diagnosed and prescribed with a HF treatment at the selected health insurance company and whose prescriptions were filled in Audifarma.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-11-16 (Actual); Study Completion 2022-11-16 (Actual)

PRIMARY OUTCOMES:
Treatment initiation patterns | Database analysis: HF patients from June 1st, 2019 to May 31st, 2020
  Treatment initiation patterns of patients with Heart Failure (HF) in an outpatient setting from Colombia.

SECONDARY OUTCOMES:
Clinical characteristics at baseline - Symptoms and signs: Dyspnea | Database analysis: HF patients from June 1st, 2019 to May 31st, 2020
Clinical characteristics at baseline - Symptoms and signs: Fatigue | Database analysis: HF patients from June 1st, 2019 to May 31st, 2020
Clinical characteristics at baseline - Symptoms and signs: Lower limb edema | Database analysis: HF patients from June 1st, 2019 to May 31st, 2020
Clinical characteristics at baseline - Laboratory data: Hemoglobin and hematocrit level | Database analysis: HF patients from June 1st, 2019 to May 31st, 2020
Clinical characteristics at baseline - Laboratory data: Left ventricular ejection fraction (LVEF) | Database analysis: HF patients from June 1st, 2019 to May 31st, 2020
Clinical characteristics at baseline - Laboratory data: EKG: main findings | Database analysis: HF patients from June 1st, 2019 to May 31st, 2020
Clinical characteristics at baseline - Laboratory data: Levels of NT-proBNP (N-terminal pro-B-type natriuretic peptide) or BNP (B-type natriuretic peptide) | Database analysis: HF patients from June 1st, 2019 to May 31st, 2020
Clinical characteristics at baseline - Laboratory data: Serum Creatinine | Database analysis: HF patients from June 1st, 2019 to May 31st, 2020
Subsequent treatment changes | Database analysis: HF patients from June 1st, 2019 to May 31st, 2020
  Determination of subsequent treatment changes in HF outpatient.
Pattern of use of HF medications according to the classification of HF by left ventricular ejection fraction: Betablockers BB | Database analysis: HF patients from June 1st, 2019 to May 31st, 2020
Pattern of use of HF medications according to the classification of HF by left ventricular ejection fraction: Angiotensin receptor blockers ARB | Database analysis: HF patients from June 1st, 2019 to May 31st, 2020
Pattern of use of HF medications according to the classification of HF by left ventricular ejection fraction: Angiotensin-converting enzyme inhibitors ACEI | Database analysis: HF patients from June 1st, 2019 to May 31st, 2020
Pattern of use of HF medications according to the classification of HF by left ventricular ejection fraction: Calcium-channel blockers CCB | Database analysis: HF patients from June 1st, 2019 to May 31st, 2020
Pattern of use of HF medications according to the classification of HF by left ventricular ejection fraction: Mineralocorticoid receptor antagonist MRA | Database analysis: HF patients from June 1st, 2019 to May 31st, 2020
Pattern of use of HF medications according to the classification of HF by left ventricular ejection fraction: Angiotensin receptor-neprilysin inhibitor ARNI | Database analysis: HF patients from June 1st, 2019 to May 31st, 2020
Pattern of use of HF medications according to the classification of HF by left ventricular ejection fraction: Sodium-glucose co-transporter 2 inhibitors SGLT2i | Database analysis: HF patients from June 1st, 2019 to May 31st, 2020

CONTACTS AND LOCATIONS:
Locations (1):
- Many Locations, Multiple Locations, Colombia

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.